## **Statistical Analysis Plan**

For

A Clinical Study Comparing the Basic Performance and Blood Compatibility Characteristics of Nipro ELISIO-H, Gambro Polyflux Revaclear and Fresenius Optiflux Dialyzers

NCT02433210

July 23, 2019

## Software:

Data were analyzed in house using SigmaPlot for Windows 11.2 (Systat Software, Inc., San Jose, CA, USA) for statistical analysis.

## Methods:

Parametric non-paired t-test was used to compare groups except where the data failed the normality test or the variance test, then the nonparametric Mann–Whitney Rank Sum was utilized to test for significance.